CLINICAL TRIAL: NCT06506227
Title: Research on Key Technologies for Risk Prediction and Precise Diagnosis and Treatment of Adolescent Idiopathic Scoliosis Based on Epigene-phenotype
Brief Title: Research on Key Technologies for Risk Prediction and Precise Diagnosis and Treatment of AIS Based on Epigene-phenotype
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-KLS-039-02
Record Dates: First submitted 2024-06-30; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-05

CONDITIONS: Adolescent Idiopathic Scoliosis
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- according to the order of their visits then were assigned numbers (Experimental): The patients were assigned numbers according to the order of their visits, and after obtaining informed consent, they were divided into a treatment group and a control group to conduct a prospective cohort study.
  Interventions: Behavioral: Low risk experimental group; Behavioral: Medium risk experimental group; Genetic: High risk experimental group; Behavioral: Control group COBB 10-20°; Behavioral: Control group COBB 20-45°; Behavioral: Control group COBB >45°; Other: Experimental group (AIS group); Other: Control group (healthy control); Other: Controlled follow-up before and after AIS
- According to the order of their visits to the clinic, given the appropriate number, (Experimental): According to the order of their visits to the clinic, given the appropriate number, divided into the test group and the control group, in strict accordance with the results of the group, the appropriate treatment and observation of the group, the teams of personnel and the implementation of clinical treatment should not be the same person.
  Interventions: Behavioral: Low risk experimental group; Behavioral: Medium risk experimental group; Genetic: High risk experimental group; Behavioral: Control group COBB 10-20°; Behavioral: Control group COBB 20-45°; Behavioral: Control group COBB >45°; Other: Experimental group (AIS group); Other: Control group (healthy control); Other: Controlled follow-up before and after AIS

INTERVENTIONS:
Behavioral: Low risk experimental group — Guiding + Manipulation + Traditional Chinese Medicine
Behavioral: Medium risk experimental group — Guiding + Manipulation + Traditional Chinese Medicine + Specific Exercise Therapy + Orthopedic Braces
Genetic: High risk experimental group — Guiding + Manipulation + Traditional Chinese Medicine + Specific Exercise Therapy + Orthopedic Braces + Specialized Inpatient Rehabilitation
Behavioral: Control group COBB 10-20° — Specific Exercise Therapy
Behavioral: Control group COBB 20-45° — Orthopedic Braces + Specific Exercise Therapy
Behavioral: Control group COBB >45° — Orthopedic Braces + Specific Exercise Therapy + Recommended Surgery
Other: Experimental group (AIS group) — Molecular marker exploration and validation
Other: Control group (healthy control) — Molecular marker exploration and validation
Other: Controlled follow-up before and after AIS — Construction and validation of AIS risk prediction model completed

SUMMARY:
Mining AIS biomarkers, elucidating the new mechanism of AIS pathogenicity, constructing risk prediction models, optimizing AIS precise diagnosis and treatment techniques, formulating precise diagnosis and treatment protocols and technical specifications for AIS combined with Chinese and Western medicine with independent intellectual property rights, and realizing the full coverage of Zhejiang Province by the end of 2026, so as to form the "Zhejiang experience" of AIS diagnosis and treatment.

DETAILED DESCRIPTION:
Currently, there are problems of high genetic and phenotypic heterogeneity in AIS research, lack of in-depth epigenetic studies, and lack of clarity in pathogenic mechanisms. This project proposes to use EWAS technology, combined with a hybrid model of multidimensional and multimodal data fusion, to realize a multi-omics joint analysis, to clarify the amount of synergistic effects between multi-omics risk factors and AIS, to draw a map of modifiable risk factors, to clarify AIS biomarkers, and to reveal AIS To clarify the biomarkers of AIS and reveal the pathogenic mechanism of AIS. Currently, the clinical diagnosis and treatment of AIS is highly subjective and lacks objective and accurate risk prediction, which makes it easy to make wrong clinical decisions, resulting in insufficient, delayed or excessive treatment, missing the optimal time for treatment, and poor clinical efficacy. This project intends to establish a multi-dimensional and multi-modal dynamic database, use the unified model construction technology, combined with the sample imbalance model, to construct a unified and accurate prediction model for AIS, to perform clinical typing and risk stratification for AIS, to establish individualized and accurate diagnostic and treatment protocols for AIS, to improve the efficacy of AIS, to obtain high-quality clinical evidence, and to formulate industry-recognized clinical prevention and treatment standards, norms, and guidelines. Through mining AIS biomarkers, elucidating new mechanisms of AIS pathogenicity, constructing risk prediction models, optimizing AIS precision diagnosis and treatment techniques, and formulating precise diagnosis and treatment protocols and technical specifications for AIS combining Chinese and Western medicine with independent intellectual property rights, the project will achieve full coverage of Zhejiang Province by the end of 2026, forming the "Zhejiang experience" in AIS diagnosis and treatment. Zhejiang experience" will be formed in AIS diagnosis and treatment. The promotion of the results can realize the precision of AIS diagnosis and treatment, improve the efficacy of AIS treatment, reduce the incidence of severe scoliosis, reduce medical expenditure by billions of dollars, and alleviate the economic burden on families and society.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with AIS;② Sex is not limited, age 10-18 years old; ③ Those who sign the informed consent and can cooperate with follow-up visits; ④ Those who can cooperate with X-ray, chemical test, genetic test and other examination and evaluation for the measurement of relevant indexes.

Exclusion Criteria:

* Subjects with spine-related diseases such as Marfan's syndrome;

  * Subjects with previous ankylosing spondylitis, spinal neurofibroma, spinal tuberculosis, spinal trauma and other spine-related diseases;

    * Subjects with combined serious medical diseases and psychiatric patients;

      * Those with ECOG score > 2, which may have an impact on the study results;

        * Those who are affected by external factors such as economy, individualized differences, etc., so that they cannot complete the study.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2000 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cobb Angle | Pre-treatment, 3, 6, 9, 12 months post-treatment
  Cobb's angle is an angle used to measure the severity of scoliosis by measuring the angle of lateral curvature to assess the degree of scoliosis.
Trunk Rotation Degree -Angle of Trunk Rotation | Pre-treatment, 3, 6, 9, 12 months post-treatment
  The patient stood with feet shoulder-width apart and bent forward with hands to palms, and the maximum degree of spinal razorback was measured with the Scoliometer Scoliosis Screening Scale.
Coronal Balance | Pre-treatment, 3, 6, 9, 12 months post-treatment
  A plumb line is usually used to determine coronal plane balance. In the coronal plane of a normal spine, a plumb line leading from the center of the C7 vertebra will pass through the center of the sacrum or within 1 cm to the left and right of the S1 spinous process.
Sagittal Balance | Pre-treatment, 3, 6, 9, 12 months post-treatment
  Sagittal Balanced descriptions in the sagittal plane are an important way to assess scoliosis and its impact on body structure and function.
Frontal Convexity Of the Spine Angle | Pre-treatment, 3, 6, 9, 12 months post-treatment
  Your doctor will ask you to stand or sit down and then take x-ray pictures of your spine from the side. These pictures show the curve and curvature of the spine, from which the doctor can assess the condition of the lordosis.
Offside Convexity Of the Spine Angle | Pre-treatment, 3, 6, 9, 12 months post-treatment
  Your doctor will ask you to stand or sit down and then take x-ray pictures of your spine from the side. These pictures clearly show the curve and curvature of the spine, and the doctor can use these images to evaluate the condition of the kyphosis.
Electromyographic (AEMG) indicators | Pre-treatment, 3, 6, 9, 12 months post-treatment
  The obtained surface EMG signal data were input into MegaWin 2.3 signal processing software to extract and analyze linear metrics (mean frequency, median frequency, muscle activity intensity, etc.), and nonlinear metrics (multi-scale sample entropy, fractal dimension, coherence, etc.)
Electroencephalographic (EEG) Index | Pre-treatment, 3, 6, 9, 12 months post-treatment
  Matlab based software and its toolkit EEGLAB were used to preprocess the data and get clean EEG signal. The effective number of channels acquired in this study was 18 leads. Fifteen 2s segments (i.e., 45s of data) were randomly selected for each subject to obtain δ (1-4Hz), θ (4-8Hz), α (8-13Hz), and β (13-30Hz), and the functional connectivity of the different bands was calculated separately.
Postural Posture Assessment | Pre-treatment, 3, 6, 9, 12 months post-treatment
  Measurements of trunk offset angle, pelvic tilt angle, thoracic lordosis angle, lumbar lordosis angle, the sum of the maximum angle of vertebral body left-right rotation, the sum of the maximum left-right deviation of the trunk, and the angle of primary bending and lateral curvature can be obtained after completion of the filming.
Balance Function | Pre-treatment, 3, 6, 9, 12 months post-treatment
  Subjects remained stationary with eyes open for 30 seconds, and four parameters of COP were recorded: area of COP oscillation, mean oscillation velocity in the anteroposterior (AP) and medial-lateral (ML) directions, and length of movement.
Questionnaire on Spinal Health of Children and Adolescents | Pre-treatment, 3, 6, 9, 12 months post-treatment
  The Spine Health Questionnaire for Children and Adolescents is designed to understand and assess the spine health status and related behaviors of this age group in their daily lives.
Skeletal maturity (Risser's sign) | Pre-treatment, 3, 6, 9, 12 months post-treatment
  Doctors determine a child's bone age based on the closest standard x-ray image in the atlas to how the child's bones appear on the x-ray.
Types of scoliosis | Pre-treatment, 3, 6, 9, 12 months post-treatment
  Although scoliosis presents all lateral curvature and vertebral rotation in the spinal phase, we can categorize it into different types based on the number of degrees of scoliosis when the degree of scoliosis is greater than ten degrees in the online screen slice mountain.
Sagittal plane axial distance (SVA) | Pre-treatment, 3, 6, 9, 12 months post-treatment
  Sagittal plane axial distance (SVA) is one of the most important indicators of spinal and body postural balance, especially when assessing anterior-posterior spinal balance. It is usually measured by imaging (e.g., X-rays or MRI) and is used to quantify the anterior-posterior positional differences between the head and a pelvis.
Muscle and bone ultrasound | Pre-treatment, 3, 6, 9, 12 months post-treatment
  Morphological characteristics of the paravertebral muscles were extracted by ultrasonography of the morphology and elasticity of the paravertebral muscles of the enrolled patients.
Number of participants with Chemical testing | Pre-treatment, 3, 6, 9, 12 months post-treatment
  Subjects were obtained for routine blood, urine, biochemistry, thyroid function, sex hormones, allergens, growth hormone, leptin, estrogen, melatonin, and other tests.
Number of participants with Blood samples | Pre-treatment, 3, 6, 9, 12 months post-treatment
  Venous blood samples were collected from all included patients at 5 mL per person.The obtained blood samples were placed at -8°C. Samples were immediately separated, partitioned and stored after collection, and some blood samples were immediately sent to the hospital for biochemical indexes.
Urine test | Pre-treatment, 3, 6, 9, 12 months post-treatment
  Drink little or no water before going to bed, and try to retain urine in the bladder for more than 4 hours, use a sterile wide-mouth container to collect, discard the anterior part of the urine, and retain about 10mL of the middle part of the urine into a sterile container, and send it to the test immediately.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Zhong, bachelor, Study Director — The First Affiliated Hospital of Zhejiang Chinese Medical University
Locations (1):
- Prokin balance apparatus, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No